CLINICAL TRIAL: NCT01168830
Title: BIOTRONIKS-Safety and Clinical Performance Of the First Drug-Eluting Generation Absorbable Metal Stent In Patients With de Novo Lesions in NatiVE Coronary Arteries (BIOSOLVE - I)
Brief Title: First in Man Trial - BIOSOLVE-I
Acronym: BIOSOLVE-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1007
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: de Novo Lesions in Native Coronary Arteries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational device (Experimental)
  Interventions: Device: AMS-3.0

INTERVENTIONS:
Device: AMS-3.0

SUMMARY:
First in Man Trial with the drug eluting absorbable metal scaffold. To assess safety

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years and < 80 years of age
* Written patient informed consent available prior to PCI
* Patients with stable or unstable angina pectoris or documented silent ischemia
* Patient eligible for PCI
* Patient acceptable candidate for coronary artery bypass surgery

Exclusion Criteria:

* Left ventricular ejection fraction of < 30%
* Presence of a visible thrombus in the target vessel visualized by angiography
* Lesion and/or way to lesion extremely calcified (e.g. IVUS catheter can not reach/cross the lesion)
* Patients with three-vessel where all three vessels require treatment
* Patients with previous CABG in the target vessel(s)
* Patients with known coronary artery spasm
* Myocardial infarction (STEMI/NSTEMI) within 4 weeks of the intended treatment. Determination of CKMB and/or troponin T or I is required.
* Patients with planned major surgery within 12 months after coronary intervention
* Patients with risk of either acetylsalicylic acid, clopidogrel or Prasugrel cessation
* Patients under current Phenprocoumon or Cumarine therapy
* Impaired renal function (serum creatinine > 2.0mg/dl or 177micromol/l, determined within 72 hours prior to intervention)
* Additional coronary lesions (restenotic or de novo) in the same vessel which requires treatment
* Totally occluded coronary artery (TIMI flow 0)
* Lesions located within arterial or venous graft
* Ostial lesions
* Previous and/or planned brachytherapy of target vessel
* Target lesion located in left main coronary artery
* Stroke or TIA < 6 months prior to procedure
* Patient with signs of a cardiogenic shock
* Surgeries of any kind within 30 days prior to screening
* Patient with bleeding diathesis in whom anticoagulation or antiplatelet medication is contraindicated
* Pregnant and/or breast-feeding females or females who intend to become pregnant
* Patient currently enrolled in other investigational device or drug trial
* Patient with expected incompliance to medical (antiplatelet, anticoagulation) therapy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure | 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (6):
- Middelheim Hospital, Antwerp, Belgium
- Germany (3):
  - Universitätsklinik Essen, Westdeutsches Herzzentrum, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Lukaskrankenhaus Neuss, Neuss
- Catharina Ziekenhuis, Eindhoven, Netherlands
- Luzerner Kantonsspital, Lucerne, Switzerland

REFERENCES:
- [Derived] Waksman R, Prati F, Bruining N, Haude M, Bose D, Kitabata H, Erne P, Verheye S, Degen H, Vermeersch P, Di Vito L, Koolen J, Erbel R. Serial observation of drug-eluting absorbable metal scaffold: multi-imaging modality assessment. Circ Cardiovasc Interv. 2013 Dec;6(6):644-53. doi: 10.1161/CIRCINTERVENTIONS.113.000693. Epub 2013 Nov 19. PMID 24254708
- [Derived] Haude M, Erbel R, Erne P, Verheye S, Degen H, Bose D, Vermeersch P, Wijnbergen I, Weissman N, Prati F, Waksman R, Koolen J. Safety and performance of the drug-eluting absorbable metal scaffold (DREAMS) in patients with de-novo coronary lesions: 12 month results of the prospective, multicentre, first-in-man BIOSOLVE-I trial. Lancet. 2013 Mar 9;381(9869):836-44. doi: 10.1016/S0140-6736(12)61765-6. PMID 23332165